CLINICAL TRIAL: NCT01045408
Title: The Adjuvant Effect of Berry Extract on Triple Therapy for Helicobacter Pylori Eradication
Brief Title: The Effect of Berry Extract on Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: HUNG,CHI-JEN, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKH-TMU-98-02
Record Dates: First submitted 2009-12-29; First posted 2010-01-11 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Increase the Eradication Rate of Helicobacter Pylori
Keywords: Helicobacter pylori; Berry extract; Triple therapy
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berry (Placebo Comparator)
  Interventions: Dietary Supplement: Berry extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Berry extract

INTERVENTIONS:
Dietary Supplement: Berry extract — Berry extract for weeks

SUMMARY:
Helicobacter pylori (HP) is the major risk factors of gastritis, gastric ulcers, duodenal ulcers, mucosa associated lymphoid tissue lymphoma and gastric cancer. Helicobacter pylori are found in 70-90% of the population in developing countries and in 25-50% of developed countries.

DETAILED DESCRIPTION:
One-week of triple therapy composed of a proton pump inhibitor plus two antibiotics is currently regarded as the gold standard for HP eradication. However, the eradication rate continues to be disappointing. Poor patient compliance and bacterial resistance are the main factors contributing to treatment failure. Therefore, it is urgently necessary to develop a non-antibiotic alternative therapy to increase the eradication rates of Helicobacter pylori. Some literatures reported that cranberry may inhibit Helicobacter pylori adhesion to the human gastric mucus and may reduce Helicobacter pylori infection in adults. The aims of his experiment were to explore the impact of berry extract on triple therapy for Helicobacter pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18

Exclusion Criteria:

* Pregnancy or breastfeeding
* Use of antibiotics 2 weeks prior to inclusion
* Previous eradication treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks after Eradication of Helicobacter pylori

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yi Huang, Ph.D, Principal Investigator — Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan